CLINICAL TRIAL: NCT02493816
Title: Phase I Study of Lentiviral-mediated COL7A1 Gene-modified Autologous Fibroblasts in Adults With Recessive Dystrophic Epidermolysis Bullosa.
Brief Title: Safety Study of Gene-modified Autologous Fibroblasts in Recessive Dystrophic Epidermolysis Bullosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LENTICOL-F
Record Dates: First submitted 2015-05-21; First posted 2015-07-10 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2018-08

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gene-modified autologous fibroblasts (Experimental): 3 intradermal injections of COL7A1 gene-modified autologous fibroblasts will be administered on day 0 only.
  Interventions: Drug: Gene-modified autologous fibroblasts

INTERVENTIONS:
Drug: Gene-modified autologous fibroblasts — 3 intradermal injections of COL7A1 gene-modified autologous fibroblasts will be administered on day 0 only.
  Other Names: COL7A1 gene-modified autologous fibroblasts

SUMMARY:
Recessive dystrophic epidermolysis bullosa (RDEB) is a severe form of blistering skin disease caused by mutations in COL7A1 gene. This study aims to assess the safety of intradermal injections of gene-modified autologous fibroblasts in 5-10 adults with RDEB.

DETAILED DESCRIPTION:
Recessive dystrophic epidermolysis bullosa (RDEB) is a severe form of blistering skin disease caused by mutations in COL7A1 gene. This study aims to assess the safety of intradermal injections of gene-modified autologous fibroblasts in 5-10 adults with RDEB.

This is an open-label single-centre phase I study with primary objective to evaluate the adverse and serious adverse events over 12 months' follow-up period. Secondary objectives include (1) analysis of type VII collagen (C7) expression and morphology of anchoring fibrils in the injected areas of the skin; (2) analysis of immune response to newly expressed C7.

Each study participant will receive three intradermal injections of COL7A1 gene-modified autologous fibroblasts on Day 0 only. Each subject will undergo an initial screening including a physical examination and assessment of disease severity. Blood analyses and skin biopsies will be performed at various time points as per the monitoring schedule over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and genetic diagnosis of RDEB with confirmed bi-allelic COL7A1 mutations.
2. A reduced number or morphologically abnormal anchoring fibrils confirmed by TEM.
3. At least 5x8cm of intact skin on the trunk and/or extremities that is suitable for cell injections.
4. Able to undergo local anaesthesia.
5. Subjects aged ≥ 17 years and able to give informed consent prior to the first study intervention.

Exclusion Criteria:

1. Subjects who received other investigational medicinal products within 6 months prior to enrolment into this study.
2. Past medical history of biopsy proven skin malignancy.
3. Subjects who have received immunotherapy including oral corticosteroids (Prednisolone >1mg/kg) for more than one week (intranasal and topical preparations are permitted) or chemotherapy within 60 days of enrolment into this study.
4. Known allergy to any of the constituents of the investigational medicinal product (IMP).
5. Subjects with BOTH:

   * positive serum antibodies to C7 confirmed by ELISA and
   * positive IIF with binding to the base of salt split skin.
6. Subjects who are pregnant or of child-bearing potential who are neither abstinent nor practising an acceptable means of contraception when this is in line with the usual and preferred lifestyle of the subject, as determined by the Investigator, for 12 months after the cell injections.
7. Subjects with positive results for HIV, Hepatitis B, Hepatitis C, HTLV or Syphilis.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs), Serious Adverse Events (SAEs), Adverse Reactions (ARs) and Serious Adverse Reactions (SARs) at each visit over 12 months' follow up period. | 12 months

SECONDARY OUTCOMES:
Type VII collagen protein expression, measured by direct immunofluorescence, in the treated and untreated skin | Week 2, Month 3 and Month 12
Morphology of anchoring fibrils, measured by transmission electron microscopy, in the treated and untreated skin | Week 2, Month 3 and Month 12
Vector copy number, measured by q-PCR, in the treated and untreated skin | Week 2, Month 3 and Month 12
Anti-type VII collagen antibodies measured by ELISA and indirect immunofluorescence | Week 2, Month 1, Month 3, Month 6 and Month 12
T-cell responses to full length type VII collagen measured by ELISPOT | Week 2, Month 1, Month 3, Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: John A McGrath, FRCP, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong T, Gammon L, Liu L, Mellerio JE, Dopping-Hepenstal PJ, Pacy J, Elia G, Jeffery R, Leigh IM, Navsaria H, McGrath JA. Potential of fibroblast cell therapy for recessive dystrophic epidermolysis bullosa. J Invest Dermatol. 2008 Sep;128(9):2179-89. doi: 10.1038/jid.2008.78. Epub 2008 Apr 3. PMID 18385758
- [Result] Lwin SM, Syed F, Di WL, Kadiyirire T, Liu L, Guy A, Petrova A, Abdul-Wahab A, Reid F, Phillips R, Elstad M, Georgiadis C, Aristodemou S, Lovell PA, McMillan JR, Mee J, Miskinyte S, Titeux M, Ozoemena L, Pramanik R, Serrano S, Rowles R, Maurin C, Orrin E, Martinez-Queipo M, Rashidghamat E, Tziotzios C, Onoufriadis A, Chen M, Chan L, Farzaneh F, Del Rio M, Tolar J, Bauer JW, Larcher F, Antoniou MN, Hovnanian A, Thrasher AJ, Mellerio JE, Qasim W, McGrath JA. Safety and early efficacy outcomes for lentiviral fibroblast gene therapy in recessive dystrophic epidermolysis bullosa. JCI Insight. 2019 Jun 6;4(11):e126243. doi: 10.1172/jci.insight.126243. eCollection 2019 Jun 6. PMID 31167965

DOCUMENTS (2):
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT02493816/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02493816/SAP_001.pdf